CLINICAL TRIAL: NCT00488657
Title: Treating Speech Disorders in Patients With Parkinson's Disease Using Altered Auditory Feedback
Brief Title: Improve Speech Using an In-the-ear Device in Parkinson's Disease
Acronym: MJFFSpeech
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Emily Wang, PhD, Rush University Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: RushUMC
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Parkinson's Disease; Dysarthria
Keywords: speech; Parkinson's disease; treatment; speech intelligibility; speaking rate
MeSH Terms: conditions — Parkinson Disease; Dysarthria; Speech; Speech Intelligibility

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): In the ear device to provide altered auditory feedback
  Interventions: Device: SpeechEasy Model ITC

INTERVENTIONS:
Device: SpeechEasy Model ITC — The delayed auditory feedback ranging from 50 to 220 ms, and the altered frequency feedback ranging from 500 to 2,000 Hz.

SUMMARY:
This project will systematically examine the therapeutic effect of altered auditory feedback provided by the in-the-ear device on the speech impairments in patients with Parkinson's disease.

Many patients with PD have difficulty starting their speech even though they know the words they want to say. They experience 'freezing' of the jaw, tongue and lips. When they eventually get their speech started, they have a hard time moving it forward. They keep on saying the same words or phrases over and over again while their voice gets softer and softer. Many words also run together. These symptoms make patients' speech very hard to understand and directly affect their care and quality of life. Currently, there is no effective medical or surgical treatment for these speech symptoms.

We have tested an in-the-ear therapeutic device that provides altered auditory feedback in eight patients with PD and moderate to severe speech impairment and the results are encouraging. We will recruit 100 patients with PD and moderate to severe speech impairment for Phase A and 20 for Phase B of the study. They will use the device routinely to provide the altered auditory feedback as they speak to improve their speech intelligibility.

DETAILED DESCRIPTION:
Speech problems are common in patients with Parkinson's disease (PD). At an early stage, patients may find it hard to project their voice. As the disease progresses, patients start to have difficulty starting their speech even though they know the words they want to say. They experience 'freezing' of the jaw, tongue and lips. When they eventually get their speech started, they have a hard time moving it forward. They keep on saying the same words or phrases over and over again while their voice gets softer and softer. Many words also run together or are slurred. These symptoms make patients' speech very hard to understand and directly affect their care and quality of life. Unfortunately, these symptoms have not responded to medication or surgery like other non-speech motor symptoms do. In fact, some surgical treatment could even make speech worse while other motor function such as walking improves. Traditional behavior therapy for these speech symptoms has not been successful either because these symptoms cannot be controlled voluntarily.

Recently, we have tested an in-the-ear therapeutic device that provides altered auditory feedback in eight patients with PD and moderate to severe speech impairment. The device is housed in a hearing aid shell, and it is programmable. Patients wore the device in one ear and heard their own speech through it after a short time delay and with a shift in pitch while they spoke. The delay ranged from 50-220 ms and their pitch shifted up or down from 500-2,000 Hz. For each patient, a specific combination of the time-delay and pitch-shift was found. Our preliminary results were encouraging. Seven of the eight PD patients made significant improvement in their speech, and they were much easier to understand when they used the device.

This project will systematically examine the therapeutic effect of altered auditory feedback provided by the in-the-ear device on the speech impairments in PD. We will recruit 100 patients with PD and moderate to severe speech impairment for Phase A and 20 for Phase B of the study. The Phase A study will be a single visit while the Phase B study will be over a one-year period while the patients use the device to provide the altered auditory feedback as they speak. Both short-term and long-term benefits of altered auditory feedback on speech will be monitored. Based on the results of our preliminary study, we expect the patients' speech will improve. We hypothesize that the use of altered auditory feedback provides salient sensory information that triggers ancillary loops to allow PD patients to initiate their speech more easily and to maintain a constant speaking rate, thus making their speech more intelligible. This project has the potential to significantly impact the quality of life for patients with PD. When PD patients can express their wants and needs and can communicate effectively with their families, caretakers and physicians, their quality of life improves.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease, presence of speech problems, native English speaker

Exclusion Criteria:

* previous brain surgery, presence of dementia or depression, profound hearing loss, previous strokes or neurological disorders/conditions other than Parkinson's disease

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
speech intelligibility | 1 year

SECONDARY OUTCOMES:
hearing changes | 1 year
speaking rate | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Emily Wang, PHD, Principal Investigator — Rush University Medical Center; Leo Verhagen, MD, PHD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States